CLINICAL TRIAL: NCT05176262
Title: A Prospective Study of the Four Food Elimination Diet for Treatment of Eosinophilic Esophagitis
Status: Active, not recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Joshua Wechsler, Attending Physician, Gatroenterology, Hepatology & Nutrition, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2011-14635
Record Dates: First submitted 2021-10-06; First posted 2022-01-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4FED Group: EoE patients recruited to this observational study will be monitored for treatment response to 4FED and treatment responders will be monitored during food reintroduction

SUMMARY:
This study is to observe the efficacy of the four food elimination diet.

DETAILED DESCRIPTION:
The goals of treatment in EoE, like for most other chronic disorders, include: 1) resolution of clinical symptoms, 2) maintenance of remission and prevention of disease relapse 3) prevention of complications such as fibrosis and strictures by maintaining histological remission 4) prevention of iatrogenic treatment related adverse reactions such as nutritional deficiencies as in dietary treatment and 5) maintenance of quality of life.

Current standard of care for the treatment of EoE include either pharmacologic modality with glucocorticosteroids (oral, or swallowed spray or slurry) or diet. Swallowed steroids are the more commonly utilized form of steroid treatment modality with histological remission rates of 50-80% of subjects. The potential drawbacks of steroid therapy include side effects such as opportunistic infections, potential suppression of the pituitary-adrenal axis with prolonged use and most important disease recurrence once the medication is discontinued.

The dietary approach is based on the hypothesis that food antigen(s) trigger eosinophilic inflammation and clinical and histological remission can be induced by identifying and excluding the causative food antigen(s). It is believed that eliminating causative food antigen(s) target the cause and thus induces long term remission. The current recommendation for treatment of EoE with diet are based on a number of retrospective and observational studies.

This prospective study eliminating the four most common (cow milk protein, wheat, egg, and soy) antigens, will primarily assess the histological response in a cohort of children and will attempt to validate the findings of the previously published retrospective study. In addition by the process of orderly and sequential reintroduction of the excluded solids the investigators will identify the different foods responsible for causing esophageal inflammation and thus disease. This study will also characterize patient demographics, symptoms and histologic changes associated with the four food elimination (4-FED) process.

Health outcomes in children and adolescents related to EoE primarily focus on symptoms and histology. This does not take into consideration the health related quality of life (HRQOL), which may be conceptualized to include physical health, mental health, social functioning, role functioning, and general health perceptions.10 HRQOL has been shown to affect patient satisfaction with and adherence to treatment, and therefore long term outcomes.

The PedsQLTM 4.0 is a, self-administered, non-preference based generic instrument. It consists of a 23-item core measure of global health-related quality of life (HRQOL). The tool includes scales of physical, emotional, social and school function and is validated for children age 2-18 years. Multiple studies have demonstrated the reliability, validity and responsiveness of this instrument in healthy children and in children with chronic diseases. Even more recently developed is the PedsQLTM Eosinophilic Esophagitis Module, a disease-specific tool that has demonstrated excellent feasibility, reliability and validity in EoE patients.

ELIGIBILITY:
Inclusion criteria:

* Patients ages 12 months-18 years
* Presence of clinical symptoms related to esophageal dysfunction such as: feeding aversion, failure to thrive, vomiting, abdominal pain, dysphagia, heartburn, and food impaction
* Histologic criteria for the diagnosis of EoE with ≥15 eosinophils per high power field from review of a total of six biopsies obtained from the distal and mid (three from each site) esophagus in subjects who were adequately pre-treated with a proton-pump inhibitor- 1mg/kg/dose twice daily, up to a maximum of 40mg or 30mg per dose depending on preparation for 6-8 weeks or had a normal 24 hour ph probe study18
* Patients who agree to 4-FED as their treatment of EoE

Exclusion criteria:

* Those patients who are on oral or swallowed steroids (prior use of steroids that was discontinued more than two months prior to enrollment does not constitute an exclusion criterion)
* Patients who are unable to tolerate the 4-FED
* Patients with concurrent eosinophilic gastroenteritis or eosinophilic colitis

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Subjects will be recruited from patients evaluated at, referred to and followed at one of the participating centers. The investigator or designee will recruit participants during clinic visits or over the phone following their diagnosis of EoE and decision of treatment
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Four Food Elimination Diet | every 6-12 months, at standard of score endoscopies
  Demonstrate the efficacy of the empiric 4-FED in inducing clinical and histological remission in children with EoE.

SECONDARY OUTCOMES:
Identifying food triggers | every 6-12 months, at standard of score endoscopies
  Identify specific foods responsible for causing disease from those who successfully respond to the 4-FED.
Allergy skin prick correlation | every 6-12 months, at standard of score endoscopies
  Determine if allergy skin prick testing identifies the same foods responsible for causing esophageal inflammation as those identified based on food challenge and histology
Determining most common and least common food trigger | every 6-12 months, at standard of score endoscopies
  Determine if cow's milk protein is the most common food antigen and soy the least common food antigen causing esophageal inflammation once foods are reintroduced back into their diet.
Food reintroduction Quality of Life measurement | every 6-12 months, at standard of score endoscopies
  Determine how the 4-FED and the elimination and reintroduction of foods affects the quality of life of patients with EoE.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua B Wechsler, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kagalwalla AF, Sentongo TA, Ritz S, Hess T, Nelson SP, Emerick KM, Melin-Aldana H, Li BU. Effect of six-food elimination diet on clinical and histologic outcomes in eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1097-102. doi: 10.1016/j.cgh.2006.05.026. Epub 2006 Jul 21. PMID 16860614
- [Background] N. G, G Y, B D, et al. A prospective clinical trial of six food elimination diet and reintroduction of causative agents in adults with eosinophilic esophagitis. Gastroenterology 2008;134:727.
- [Background] Gonsalves N, Yang GY, Doerfler B, Ritz S, Ditto AM, Hirano I. Elimination diet effectively treats eosinophilic esophagitis in adults; food reintroduction identifies causative factors. Gastroenterology. 2012 Jun;142(7):1451-9.e1; quiz e14-5. doi: 10.1053/j.gastro.2012.03.001. Epub 2012 Mar 3. PMID 22391333
- [Background] Kagalwalla AF, Shah A, Li BU, Sentongo TA, Ritz S, Manuel-Rubio M, Jacques K, Wang D, Melin-Aldana H, Nelson SP. Identification of specific foods responsible for inflammation in children with eosinophilic esophagitis successfully treated with empiric elimination diet. J Pediatr Gastroenterol Nutr. 2011 Aug;53(2):145-9. doi: 10.1097/MPG.0b013e31821cf503. PMID 21788754
- [Background] Kelly KJ, Lazenby AJ, Rowe PC, Yardley JH, Perman JA, Sampson HA. Eosinophilic esophagitis attributed to gastroesophageal reflux: improvement with an amino acid-based formula. Gastroenterology. 1995 Nov;109(5):1503-12. doi: 10.1016/0016-5085(95)90637-1. PMID 7557132
- [Background] Liacouras CA, Spergel JM, Ruchelli E, Verma R, Mascarenhas M, Semeao E, Flick J, Kelly J, Brown-Whitehorn T, Mamula P, Markowitz JE. Eosinophilic esophagitis: a 10-year experience in 381 children. Clin Gastroenterol Hepatol. 2005 Dec;3(12):1198-206. doi: 10.1016/s1542-3565(05)00885-2. PMID 16361045
- [Background] Markowitz JE, Spergel JM, Ruchelli E, Liacouras CA. Elemental diet is an effective treatment for eosinophilic esophagitis in children and adolescents. Am J Gastroenterol. 2003 Apr;98(4):777-82. doi: 10.1111/j.1572-0241.2003.07390.x. PMID 12738455
- [Background] Spergel JM, Andrews T, Brown-Whitehorn TF, Beausoleil JL, Liacouras CA. Treatment of eosinophilic esophagitis with specific food elimination diet directed by a combination of skin prick and patch tests. Ann Allergy Asthma Immunol. 2005 Oct;95(4):336-43. doi: 10.1016/S1081-1206(10)61151-9. PMID 16279563
- [Background] Furuta GT, Liacouras CA, Collins MH, Gupta SK, Justinich C, Putnam PE, Bonis P, Hassall E, Straumann A, Rothenberg ME; First International Gastrointestinal Eosinophil Research Symposium (FIGERS) Subcommittees. Eosinophilic esophagitis in children and adults: a systematic review and consensus recommendations for diagnosis and treatment. Gastroenterology. 2007 Oct;133(4):1342-63. doi: 10.1053/j.gastro.2007.08.017. Epub 2007 Aug 8. PMID 17919504
- [Background] Eiser C. Children's quality of life measures. Arch Dis Child. 1997 Oct;77(4):350-4. doi: 10.1136/adc.77.4.350. No abstract available. PMID 9389244
- [Background] Carballo E, Cadarso-Suarez C, Carrera I, Fraga J, de la Fuente J, Ocampo A, Ojea R, Prieto A. Assessing relationships between health-related quality of life and adherence to antiretroviral therapy. Qual Life Res. 2004 Apr;13(3):587-99. doi: 10.1023/B:QURE.0000021315.93360.8b. PMID 15130023
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Varni JW, Seid M, Smith Knight T, Burwinkle T, Brown J, Szer IS. The PedsQL in pediatric rheumatology: reliability, validity, and responsiveness of the Pediatric Quality of Life Inventory Generic Core Scales and Rheumatology Module. Arthritis Rheum. 2002 Mar;46(3):714-25. doi: 10.1002/art.10095. PMID 11920407
- [Background] Franciosi JP, Hommel KA, DeBrosse CW, Greenberg AB, Greenler AJ, Abonia JP, Rothenberg ME, Varni JW. Development of a validated patient-reported symptom metric for pediatric eosinophilic esophagitis: qualitative methods. BMC Gastroenterol. 2011 Nov 18;11:126. doi: 10.1186/1471-230X-11-126. PMID 22099448
- [Background] Franciosi JP, Hommel KA, Greenberg AB, DeBrosse CW, Greenler AJ, Abonia JP, Rothenberg ME, Varni JW. Development of the Pediatric Quality of Life Inventory Eosinophilic Esophagitis module items: qualitative methods. BMC Gastroenterol. 2012 Sep 25;12:135. doi: 10.1186/1471-230X-12-135. PMID 23009120
- [Background] Franciosi JP, Hommel KA, Bendo CB, King EC, Collins MH, Eby MD, Marsolo K, Abonia JP, von Tiehl KF, Putnam PE, Greenler AJ, Greenberg AB, Bryson RA, Davis CM, Olive AP, Gupta SK, Erwin EA, Klinnert MD, Spergel JM, Denham JM, Furuta GT, Rothenberg ME, Varni JW. PedsQL eosinophilic esophagitis module: feasibility, reliability, and validity. J Pediatr Gastroenterol Nutr. 2013 Jul;57(1):57-66. doi: 10.1097/MPG.0b013e31828f1fd2. PMID 23478422
- [Background] Liacouras CA, Furuta GT, Hirano I, Atkins D, Attwood SE, Bonis PA, Burks AW, Chehade M, Collins MH, Dellon ES, Dohil R, Falk GW, Gonsalves N, Gupta SK, Katzka DA, Lucendo AJ, Markowitz JE, Noel RJ, Odze RD, Putnam PE, Richter JE, Romero Y, Ruchelli E, Sampson HA, Schoepfer A, Shaheen NJ, Sicherer SH, Spechler S, Spergel JM, Straumann A, Wershil BK, Rothenberg ME, Aceves SS. Eosinophilic esophagitis: updated consensus recommendations for children and adults. J Allergy Clin Immunol. 2011 Jul;128(1):3-20.e6; quiz 21-2. doi: 10.1016/j.jaci.2011.02.040. Epub 2011 Apr 7. PMID 21477849